## **Empowering Students Project**

## NCT05511298

August 16, 2022

## **Statistical Analysis Plan**

Each participant will have two observations for each primary outcome, one at pre-test and one at post-test. Because these are non-independent matched data, analyses will use a within-person design.

RQ1) Do participants experience improvement in targeted outcomes from before to after participation in the YRE program?

RQ1 will be analyzed using a paired samples t-test to determine whether post-test scores significantly differ from pre-test scores on a within-person basis. In other words, did each participant improve in the outcome domain compared to their own pre-test level.

RQ2) Do students who receive the YRE program in a traditional school setting experience a different amount of change than the students who receive the program in a non-traditional school setting?

RQ2 adds school setting (traditional vs. nontraditional) as a between-subjects variable and thus will be analyzed using a two-way mixed ANOVA. This analysis tests for an interaction between change over time and school setting, indicating whether there is differential change in outcomes from pre-test to post-test in the two school settings.